CLINICAL TRIAL: NCT03093467
Title: Effectiveness of an Internet-based Intervention for the Treatment of Depression: Towards the Improvement of the Management of Depression
Brief Title: Effectiveness of an Internet-based Intervention for the Treatment of Depression
Acronym: ASCENSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Milenio para Investigación en Depresión y Personalidad (Other)
Collaborators: Psicomedica Clinical & Research Group, Chile (Unknown); University Hospital Heidelberg (Other); National Fund for Research and Development in Health, Chile (Other)
Responsible Party: Principal Investigator, Álvaro Carrasco, Researcher, Instituto Milenio para Investigación en Depresión y Personalidad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA16I0173
Record Dates: First submitted 2017-03-14; First posted 2017-03-28 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Depression
Keywords: Internet; Mental Health
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Antidepressive Agents; Anti-Anxiety Agents; Antipsychotic Agents; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Open randomized controlled trial in one mental health center.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants receive psychiatric treatment and psychotherapy as usual. In addition, participants have access to the internet-based program ASCENSO: an adjunct support and monitoring system for the treatment of depression.
  Interventions: Behavioral: ASCENSO; Drug: Antidepressants or in combination with anxiolytics, neuroleptics or mood stabilizers.; Behavioral: Psychotherapy
- Control (Active Comparator): Patients receive psychiatric treatment and psychotherapy as usual.
  Interventions: Drug: Antidepressants or in combination with anxiolytics, neuroleptics or mood stabilizers.; Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: ASCENSO — Internet-based program: an adjunct support and monitoring system for the treatment of depression.
  Other Names: Internet-based program
  Arms: Experimental
Drug: Antidepressants or in combination with anxiolytics, neuroleptics or mood stabilizers. — Usual psychiatric treatment which may include drugs: antidepressant monotherapy or antidepressants in combination with anxiolytics, neuroleptics or mood stabilizers as needed, according to the psychiatric evaluation. Monthly controls during 5 months in average.
  Other Names: Psychiatric treatment
Behavioral: Psychotherapy — Usual treatment: brief psychotherapy. One session per week, a total of 9 sessions in average.

SUMMARY:
Depression is a highly prevalent disorder in Chile, generating important personal and social costs. This study aims to evaluate the effectiveness of the internet-based program ASCENSO as an adjunct intervention for the treatment of depression. ASCENSO provides information to promote patients' self-care, it monitors reported depression symptoms providing automatized feedback and provides the possibility of booking a counseling session via chat or by phone. To evaluate the effectiveness of ASCENSO, an open, evaluator-blind, prospective, parallel-group (one intervention group and one active control group) randomized controlled trial will be implemented in one mental health center in Santiago of Chile. The sample will be composed of adults initiating treatment for depression, and who have internet access. Participants will be randomly assigned to one of the two study arms. Randomization will be stratified by the number of patients´ previous episodes (dichotomized into none, 1 or more), following a permuted block randomization procedure. Patients in the experimental group (n=100) will receive the usual treatment plus access to the ASCENSO program. The control group (n=100) will only receive the usual treatment. At recruitment, months 6 and 9, patients' self-reported depression symptoms and quality of life will be assessed. Additionally, adherence to treatment in terms of patients' attendance to medical controls and psychotherapy sessions will be registered for both research groups.

DETAILED DESCRIPTION:
The public health system has established policies and priorities to provide access to depression treatment and to improve the quality of those services. The acknowledgment of the complexity and chronicity of the disorder has motivated the design and implementation of comprehensive disease management strategies for depression. There are experiences that show that information technologies can help to optimize the management of depression. If ASCENSO is effective, it could be a useful resource to include to the mental health services for depression in Chile.

The components of the ASCENSO program are:

Emergency. Standard Information on what to do and who to contact in a crisis situation.

Online or phone counseling. Patients can schedule a 30-minute session with a psychologist, which is conducted in a private text chatroom or over the phone.

Monitoring. Patients receive a bi-weekly email with a link to the monitoring questionnaire and automatized tailored feedback message. If a participant reports severe impairment, the ASCENSO administrator receives an alert notification and then contacts the patient.

Self-care information and blog. Web pages with basic information about depression and self-care recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depression disorder
* Internet access

Exclusion Criteria:

* previous suicide attempt
* hospitalization for a previous depressive episode
* a history of psychotic symptoms
* bipolar disorder
* organic brain disorders
* any serious disorders related to substance abuse or dependence
* antisocial personality disorder
* a serious medical condition or severe cognitive impairment
* lack of knowledge of the Spanish language
* illiteracy
* refusal or revocation of patient consent.

Patients will be evaluated using the MINI International Neuropsychiatric interview, Spanish for Chile Translation Version 6.0.0.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Change in depressivity assessed with the Beck's Depression Inventory I (BDI-I) | Baseline, months 6 and 9.
  Beck's Depression Inventory I (BDI-I) total score (score range 0 - 63)

SECONDARY OUTCOMES:
Change in quality of life change assessed with the EuroQol/EQ-5D | Baseline, months 6 and 9.
  EuroQol/EQ-5D (EQ-index range 0 - 1)

OTHER OUTCOMES:
Number of attended and missed treatment appointments | Months 6 and 9.
  Adherence to treatment in terms of patients' attendance to medical controls and psychotherapy sessions.
Number of patients that dropout from treatment | Months 6 and 9.
  Number of patients that dropout from psychiatric or psychotherapeutic treatment during the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro E. Carrasco, PhD, Principal Investigator — Millennium institute for research on depression and personality (MIDAP); Janet C. Pérez, PhD, Principal Investigator — Millennium institute for research on depression and personality (MIDAP)
Locations (1):
- Psicomedica, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Yes
Individual quantitative participant data that underlie the reported results, after deidentification (text, tables and figures).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: These data will be available to researchers who provide a methodologically sound proposal for the purposes of achieving specific aims outlined in that proposal. Proposals should be directed to J. Carola Pérez via email (janetperez@udd.cl) or Olga Fernandez (mofernandez36@gmail.com) and will be reviewed by both researchers. Requests to access data to undertake hypothesis-driven research will not be unreasonably withheld. To gain access, data requesters will need to sign a data access agreement and to confirm that data will only be used for the agreed purpose for which access was granted and this these data will be not shared to other people.

REFERENCES:
- [Background] Alvarado R, Rojas G. [Evaluation of the program for detection and treatment of depression in Chilean primary health care centers]. Rev Med Chil. 2011 May;139(5):592-9. Epub 2011 Sep 16. Spanish. PMID 22051709
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Espinosa HD, Carrasco A, Moessner M, Caceres C, Gloger S, Rojas G, Perez JC, Vanegas J, Bauer S, Krause M. Acceptability Study of "Ascenso": An Online Program for Monitoring and Supporting Patients with Depression in Chile. Telemed J E Health. 2016 Jul;22(7):577-83. doi: 10.1089/tmj.2015.0124. Epub 2016 Jan 7. PMID 26741190
- [Background] Fritsch R, Araya R, Solis J, Montt E, Pilowsky D, Rojas G. [A randomized trial of pharmacotherapy with telephone monitoring to improve treatment of depression in primary care in Santiago, Chile]. Rev Med Chil. 2007 May;135(5):587-95. Epub 2007 Jul 9. Spanish. PMID 17657327
- [Background] Hamine S, Gerth-Guyette E, Faulx D, Green BB, Ginsburg AS. Impact of mHealth chronic disease management on treatment adherence and patient outcomes: a systematic review. J Med Internet Res. 2015 Feb 24;17(2):e52. doi: 10.2196/jmir.3951. PMID 25803266
- [Background] Kordy H, Wolf M, Aulich K, Burgy M, Hegerl U, Husing J, Puschner B, Rummel-Kluge C, Vedder H, Backenstrass M. Internet-Delivered Disease Management for Recurrent Depression: A Multicenter Randomized Controlled Trial. Psychother Psychosom. 2016;85(2):91-8. doi: 10.1159/000441951. Epub 2016 Jan 26. PMID 26808817
- [Background] Neumeyer-Gromen A, Lampert T, Stark K, Kallischnigg G. Disease management programs for depression: a systematic review and meta-analysis of randomized controlled trials. Med Care. 2004 Dec;42(12):1211-21. doi: 10.1097/00005650-200412000-00008. PMID 15550801
- [Derived] Perez JC, Fernandez O, Caceres C, Carrasco AE, Moessner M, Bauer S, Espinosa-Duque D, Gloger S, Krause M. An Adjunctive Internet-Based Intervention to Enhance Treatment for Depression in Adults: Randomized Controlled Trial. JMIR Ment Health. 2021 Dec 16;8(12):e26814. doi: 10.2196/26814. PMID 34927594
- See also: Mental health clinic. Recruitment center. — http://ww3.psicomedica.cl/
- See also: Millennium Institute for research on depression and personality — http://midap.org
- See also: Center for psychotherapy research, Heidelberg University Hospital — http://psyres.de/
- See also: Fund for research and development in health — http://www.conicyt.cl/fonis/